CLINICAL TRIAL: NCT05588778
Title: CEREBRO - Cognitive Enhancement and Risk-reduction Through Exercise for Brain-Related Outcomes
Brief Title: Cognitive Enhancement and Risk-reduction Through Exercise for Brain-Related Outcomes
Acronym: CEREBRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, David Xavier Marquez, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3U48DP006392-04S6 (NIH)
Record Dates: First submitted 2022-10-13; First posted 2022-10-20 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Aging
Keywords: Latino; older adults; cognition; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Conduct a 6-month RCT comparing BAILAMOS™ @home/en casa and ¡En Forma y Fuerte! @home/en casa among 100 older Latino adults with symptoms of cognitive decline.
Who Masked: Participant
Masking Description: Participants will not be explicitly told which condition they are randomized to, but are likely to know. All data collectors will be blinded to participants' study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAILAMOS™ @home/en casa (Experimental): The BAILAMOS™ @home/en casa dance program is provided twice weekly for 24 weeks. Each month a new dance style is introduced by a professional dance instructor.
  Interventions: Behavioral: ¡En Forma y Fuerte! @home/en casa
- ¡En Forma y Fuerte! @home/en casa (Experimental): ¡En Forma y Fuerte! @home/en casa is an exercise and health education program designed to improve arthritis-related outcomes. The classes will meet two times per week for 90 min each for 12 weeks. Each class session consists of 60 min of exercise (flexibility, aerobics and strength training) and 30 minutes of health education using group problem solving based on SCT.
  Interventions: Behavioral: ¡En Forma y Fuerte! @home/en casa

INTERVENTIONS:
Behavioral: BAILAMOS™ @home/en casa — The BAILAMOS™ dance program and dance manual. BAILAMOS™ originally encompassed four dance styles: Merengue, Cha Cha Cha, Bachata, and Salsa. These four styles of Latin dance are generally considered the most popular in terms of recognition and preference. We have added two styles to appeal to the largely Mexican-origin Latinos in Chicago (i.e., Cumbia and Samba). The dances were jointly choreographed by the PI and Mr. Mendez, a professional dance instructor and owner of The Dance Academy of Salsa and http://www.salsachicago.com/. The PI and dance instructor co-developed the extensive manual is used by program instructors and includes background information on the authors, an introduction describing the goals of the program, and descriptions of the various styles of dance. The manual also has photos and descriptions of each dance broken down into its component parts.
  Other Names: BAILAMOS™
Behavioral: ¡En Forma y Fuerte! @home/en casa — The ¡En Forma y Fuerte! Program. ¡En Forma y Fuerte! is designed to be delivered in Spanish by bilingual, bicultural, qualified exercise instructors. Instructors are required to have an exercise instructor/specialist certification through a national organization such as the American College of Sports Medicine, American Council on Exercise, or Aerobics and Fitness Association of America, or to have an undergraduate degree in an exercise science related field. The 8 hour training uses both didactic and hands-on role modeling for delivering both the exercise and health education components of the program. Instructors in the online version will also participate in a 60 minute training designed for this new version of the program. We have previously developed an asynchronous, online instructor training for the customary program and will translate it to Spanish for this proposal.
  Other Names: Fit & Strong!

SUMMARY:
As the population ages, it is also growing more diverse. Twelve percent of older Latinos are currently diagnosed with Alzheimer's disease (AD), and it is estimated that the number of Latinos with AD will increase by 832% by 2060. Pharmacological treatments available for cognitive decline/ADRD have shown limited effectiveness in reducing cognitive and functional decline. Evidence suggests that protective factors for AD include regular physical activity (PA). Unfortunately, older Latinos are 46% less likely to engage in leisure time PA than older non-Latino whites. The investigators propose that indoor PA programs can overcome the biggest barriers to participation. Marquez and colleagues created a Spanish-language, Latin dance program (BAILAMOS™ - Balance and Activity In Latinos, Addressing Mobility in Older Adults). Smaller studies of BAILAMOS™ have found greater improvement in global cognition in the dance group compared to a health education group, and increases in brain functional connectivity. UIC faculty have also designed and tested Fit & Strong!, a PA program for older adults with arthritis, that is recognized by the National Council on Aging as an Evidence-based program and have established the feasibility of ¡En Forma y Fuerte!, an adaptation of Fit & Strong! for Latinos with arthritis. A small trial found significant improvements in lower-extremity strength, perceived physical function, and pain from baseline to 8 weeks (p < .05) that were maintained at 6 months. No major program adaptations (other than language) were observed or reported; however, the instructors provided several suggestions for program improvements, including adjusting the literacy level and length of the program. The current pandemic allows the investigators to adapt both of these evidence informed programs, the BAILAMOS™ dance program and ¡En Forma y Fuerte!, for remote delivery among older Latinos (i.e., BAILAMOS™ @home/en casa and ¡En Forma y Fuerte! @home/en casa). The overall purpose is to implement promising, evidence-informed interventions and solutions to reduce risk for ADRD and improve quality of life for persons with symptoms of cognitive decline.

DETAILED DESCRIPTION:
By 2065, the Latino population in the U.S. is expected to grow to 107 million. Currently, 12% of older Latinos are diagnosed with Alzheimer's disease (AD); it is estimated their number will increase by 832% by 2060. Latinos have a greater risk of developing chronic conditions involving modifiable lifestyle factors, and evidence suggests that cardiovascular disease risk factors may also be a risk for AD and related dementias (ADRD), thus placing Latinos at even greater risk for ADRD.

Pharmacological treatments available for ADRD have shown limited effectiveness in reducing cognitive and functional decline, thus, the establishment of interventions that can reduce ADRD risk is critical. While there is no cure for AD, evidence suggests that protective factors for AD include regular physical activity (PA). Unfortunately, older Latinos are 46% less likely to engage in leisure time PA than older non-Latino whites.

Walking and dancing are the two most commonly reported forms of PA among older Latinos. However, urban older Latinos cite unsafe neighborhoods and extreme weather conditions as significant barriers to walking. Older Latinos value functional independence, and relate physical fitness to feeling healthy and being able to perform normal activities with ease, but have rarely had traditional exercise programs adapted to their needs. The investigators propose that indoor PA programs can overcome the biggest barriers to participation. Latin dance is a particularly promising PA modality that is a culturally acceptable type of PA for middle- aged and older Latinos. Randomized controlled trials (RCTs) have examined changes in cognitive performance among several types of dance styles and have found improvements in global cognition, executive function, episodic and working memory, and attention. However, PA interventions have not implemented dance programs specifically for Latinos, a historically excluded population at high risk of cognitive impairment. Given the need to address health inequities in Latinos, Marquez and colleagues created a Spanish-language, Latin dance program (BAILAMOS™ - Balance and Activity In Latinos, Addressing Mobility in Older Adults). Smaller studies of BAILAMOS™ have found greater improvement in global cognition in the dance group compared to a health education group, and increases in brain functional connectivity. Moreover, the investigators established the feasibility and impact on PA in older Latinos who already had MCI (n=20).

UIC faculty have also designed and tested Fit & Strong!, a PA program for older adults with arthritis, that is recognized by the National Council on Aging as an Evidence-based program and have established the feasibility of ¡En Forma y Fuerte!, an adaptation of Fit & Strong! for Latinos with arthritis. A small trial found significant improvements in lower-extremity strength, perceived physical function, and pain from baseline to 8 weeks (p < .05) that were maintained at 6 months. No major program adaptations (other than language) were observed or reported; however, the instructors provided several suggestions for program improvements, including adjusting the literacy level and length of the program.

The current pandemic allows the investigators to adapt both of these evidence informed programs, the BAILAMOS™ dance program and ¡En Forma y Fuerte!, for remote delivery among older Latinos (i.e., BAILAMOS™ @home/en casa and ¡En Forma y Fuerte! @home/en casa). The overall purpose is to implement promising, evidence-informed interventions and solutions to reduce risk for ADRD and improve quality of life for persons with symptoms of cognitive decline. Our previous engagement as a collaborating center of the CDC Healthy Aging Research Network (HAN) and the CDC Healthy Brain Research Network (HBRN), plus our evidence-the focus of our NIA Roybal Center on PA and cognition, make the UIC PRC DRRRN well suited to contribute expertise to the network.

ELIGIBILITY:
Inclusion criteria include:

1. age > 60 years old;
2. self-identification as Latino/Hispanic;
3. ability to speak Spanish;
4. participation in <1 day/week of aerobic exercise;
5. mild cognitive impairment indicated by scores on the Montreal Cognitive Assessment (MoCA) of > 16 and < 25 or subjective memory complaints determined by a response of "Very often," "Often," or "Sometimes" (not "Rarely" or "Never") to the following question of the Rush Alzheimer's Disease Center: About how often do you have trouble remembering things?;
6. danced < 2 times/month over the past 12 months;
7. willingness to be randomly assigned to either study group;
8. no plans to leave the country for more than two consecutive weeks over the next 6 months.

Exclusion criteria include:

needing a caregiver for daily functioning, self-reported presence of uncontrolled cardiovascular disease or uncontrolled diabetes mellitus, pacemaker in situ, stroke, severe chronic obstructive pulmonary disease (COPD), and recent healing or unhealed fracture(s).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment and retention | Pre-intervention through study completion, an average of 1 year
  "Feasible" will entail a total of 100 participants enrolled and ≥75% retained (operationalized as take part in post-intervention testing) at year 2 end.
Feasibility - Intervention adherence | Pre-intervention through study completion, an average of 1 year
  "Feasible" will entail ≥75% participants with ≥80% of intervention sessions completed across waves.

SECONDARY OUTCOMES:
Self-Report Physical activity | Pre-intervention through study completion, an average of 1 year
  The CHAMPS Physical Activity Questionnaire for Older Adults is a change-sensitive PA scale that assesses weekly frequency and duration of lifestyle PA (leisure time, household, occupational, and transportation PA) typically undertaken by older adults.
Device-assessed Physical activity | Pre-intervention through study completion, an average of 1 year
  ActiGraph Model GT3X-Plus accelerometers (The Actigraph, Pensacola, FL) are small and lightweight triaxial accelerometers that measure accelerations in three planes. Time spent in light, moderate or vigorous intensity PA (Miller et al. cutpoints for older adults) will be assessed. Data will be included in analysis if the accelerometer displays at least 10 hours of data (> 0 count values for each hour) in a 24-hour period on at least 4 days.
Cognition | Pre-intervention through study completion, an average of 1 year
  Neuropsychological measures of executive function, attention, episodic memory, processing speed and working memory from the NIH Toolbox for the Assessment of Neurological Behavior and Function Cognition Battery (NIHTB-CB) will be used.
Health Related Quality of life | Pre-intervention through study completion, an average of 1 year
  The SF-12 scale consists of 12 items and eight scales: physical functioning (PF), role limitations due to physical problems (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and perceived mental health (MH). The composite physical (PCS) and mental health (MCS) scores are computed using the scores of the 12 items, ranging from 0 to 100, where zero reflects the lowest health level and 100 the highest level.
Social connectedness | Pre-intervention through study completion, an average of 1 year
  Social connectedness will be assessed with Cohen's Social Network Index. It is a 12-item questionnaire that assesses participation in 12 types of social relationships including spouse, parents, friends, family members, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No